CLINICAL TRIAL: NCT07266740
Title: PURSUIT: A Technologically Augmented School-based Program to Improve Child Coping and Prevent Substance Use.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Natoshia Cunningham, Associate Professor, Michigan State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00011346; G-2404-153994 (Other Grant/Funding Number: Michigan Health Endowment Fund)
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Pain; Anxiety; Mood; Stress; Feasibility Studies; Acceptability; Health Promotion; Online Mental Health Program
Keywords: Cognitive-behavioral; School; Pediatrics; Stress; Pain; Anxiety; Mood; Substance use
MeSH Terms: conditions — Anxiety Disorders; Pain; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: All youth enrolled in the study will be given access to the online self-management platform.
Masking Description: Masking does not apply to this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PURSUIT Self-Management Portal (Experimental): All youth enrolled in the study will have access to an online self-management platform, hosted by the Computerized Intervention Authoring System (CIAS). The self-management platform comprises evidence-based cognitive-behavioral psycho-education and skills broadly applicable to physical (pain) and mental (stress, mood) health symptoms. Youth aged twelve and older will have access to content related to preventing substance use. Materials include instructional videos, handouts, and worksheets.
  Interventions: Behavioral: PURSUIT

INTERVENTIONS:
Behavioral: PURSUIT — PURSUIT is an online self-management platform for youth aged 8-18 and one caregiver that provides cognitive-behavioral coping skills for physical and mental health symptoms, plus substance use prevention content for youth aged 12 and older.

SUMMARY:
The study investigators aim to test an online support platform for Michigan youth aged 8-18 years enrolled in elementary, middle, or high school and their parent/caregiver. The online support platform will be hosted on the Computerized Intervention Authoring System (CIAS) 3.0 and will provide evidence-based cognitive behavioral coping skills for physical (pain) and mental (stress, mood) health symptoms, with additional substance use prevention content for youth aged 12 and older. Evaluations will occur at baseline and then a post assessment approximately 8 weeks later.

DETAILED DESCRIPTION:
The study investigator's aims are to:

1. Evaluate the feasibility and acceptability of the PURSUIT online support platform using mixed methods.
2. Explore the impact of PURSUIT on youth's physical (pain) and mental health (stress, anxiety, mood, perceived risk of substance use) symptoms at post assessment.

Consented youth will complete a baseline assessment (week 1), and then will use the PURSUIT online platform (expected duration is 6 week), and complete a post assessment (week 8).

Within the PURSUIT platform, all youth will have access to tools teaching cognitive-behavioral strategies for managing mood, anxiety, stress, and physical pain. Youth aged 12 and older will have access to additional content presenting cognitive-behavioral strategies for reducing the risk of substance use.

Youth will provide data on their symptoms (e.g thoughts, mood, behaviors, sleep, pain, and stress) at baseline and post assessment. A caregiver will report on the child's demographics, adverse childhood experience (ACE) exposure, school performance/attendance and their own mood. At post-assessment, the youth will also be asked to take part in a brief, semi-structured interview regarding their experiences with PURSUIT.

ELIGIBILITY:
Inclusion Criteria:

* Aged eight to 18 years
* Enrolled in a Michigan elementary, middle, or high school

Exclusion Criteria:

* Age under 8
* Age over 18 years
* Non-enrollment in A Michigan school.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
PURSUIT Feasibility-Youth Retention | From baseline to post assessment, approximately 8 weeks
  The percentage of youth who complete a post-assessment measure, relative to those who complete a baseline assessment.
PURSUIT Feasibility/Acceptability | From baseline to post-assessment, approximately 8 weeks.
  Youth will complete a brief, semi-structured interview following a six-week period of engagement with the online self-management portal to assess the feasibility ("Do you think you will be able to integrate these skills into your schedule with school/work?") and acceptability of PURSUIT.

SECONDARY OUTCOMES:
Changes in pain, as measured by the Pain Visual Analog Scale (VAS) | From baseline to post-assessment, approximately 8 weeks.
  Youth will report their average pain intensity over the past two weeks using a Visual Analog Scale (VAS). Responses range from 0 (no pain) to 10 (worst imaginable pain), with ratings ≥ 3 indicating moderate pain.
Change in functional disability, measured using the Functional Disability Inventory (FDI) | From baseline to post-assessment, approximately 8 weeks.
  The 15-item FDI assesses youths' difficulty performing tasks across home, school, recreational, and social settings over the "past few days" due to physical symptoms. Items are rated from 0 ("no trouble") to 4 ("impossible") and summed, yielding total scores of 0-60 with scores ≥7 suggesting greater than minimal disability
Changes in post-traumatic stress disorder symptoms (PTSD), measured using the UCLA Reaction Index for DSM-5 Brief Screening Form | From baseline to post-assessment, approximately 8 weeks.
  The UCLA Reaction Index for DSM-5 Brief Screening Form is an 11-item measure of how often youth experienced psychological stress and physiological reactivity due to internal or external trauma reminders, intrusive trauma-related memories, avoidance of internal and external reminders of trauma, emotional dysregulation, attention issues, feelings of detachment, and sleep disturbance over the past month. Items are scored from zero (none of the time) to four (most of the time) and summed; scores of 11-20 suggest mild PTSD symptoms, while scores ≥21 are indicative of potential PTSD. We adapted this measure to not query the type of traumatic exposure experienced by youth. It will only be completed by those who endorse exposure (yes/no) to a frightening or upsetting event.
Change in anxiety symptoms, measured using the Screen for Child Anxiety Related Disorders (SCARED) | From baseline to post-assessment, approximately 8 weeks.
  The 41-item Screen for Child Anxiety Related Disorders (SCARED) assesses past 3-month anxiety symptoms. Items are scored on a 3-point Likert-style scale (0 = not true or hardly ever true, 2=very true or often true), and summed to yield total scores of 0-82 with higher scores indicating greater anxiety and scores ≥25 suggesting clinical significance.
Change in depressive symptoms, measured using the PROMIS Pediatric Short Form 8a | From baseline to post-assessment, approximately 8 weeks.
  Youth will report the frequency (1=never, 5=almost always) of past-week depressive symptoms (e.g., sadness, loneliness) using the eight-item PROMIS Pediatric Depressive Symptoms Short Form 8a. Raw summed scores (range 8 to 40) are converted to T-scores (mean 50, standard deviation 10), with T-scores >55 suggesting mild or higher symptoms.
Change in fatigue symptoms; as measured by the PROMIS Pediatric Short Form 10a | From baseline to post-assessment, approximately 8 weeks.
  Past week fatigue symptoms will be self-reported by youth using the 10-item PROMIS Pediatric Short Form. Items ("Being tired made it hard for me to play or go out with my friends as much as I'd like") are rated on a 5-point Likert-style scale (1=never, 5=almost always) and summed in to total scores, which are converted into T-scores (>55 suggesting at least mild symptoms).
Change in sleep disturbance symptoms, measured using the PROMIS Pediatric Sleep Disturbance Short Form 8a | From baseline to post-assessment; approximately 8 weeks
  The frequency (1=never, 5=almost always) with which youth experienced sleep disturbance symptoms (e.g., trouble falling or staying asleep) in the past week will be assessed using the eight-item PROMIS Pediatric Sleep Disturbance Short Form. T-scores (>55 indicative of mild or greater symptoms) will be derived from summed raw scores.
Change in youths' perceived risk of substance use; measured using Monitoring The Future items | From baseline through post-assessment; approximately 8 weeks.
  Youth age 12 and older will report how risky (1= No Risk, 4=Great Risk) they perceive different cigarette, cannabis, alcohol, or vaping use behaviors (e.g., occasional versus regular use) using 12 items from the 2023 Monitoring the Future (MTF) study. MTF is an ongoing longitudinal panel study conducted by the University of Michigan that includes annual surveys of nationally representative samples of 8th, 10,th and 12th grade youth.
Change in youth's substance use behaviors; assessed using the Screening to Brief Intervention (S2B1) | From baseline through post-assessment; approximately 8 weeks.
  The frequency (never, once or twice, monthly, weekly or more often) of past-year nicotine, alcohol, cannabis, and other substance use behaviors will be assessed for youth 12 years and older using the youth-reported Screening to Brief Intervention (S2BI)
Changes in caregivers' depression, anxiety, and stress as measured by the Depression Anxiety and Stress Scales 21 (DASS21) | From baseline to post-assessment, approximately 8 weeks.
  The DASS21 depression, anxiety, and stress on a scale of 0-63 with 0 indicating low levels of these feelings, and 63 indicating high levels. This measure will only be completed by caregivers.
Change in stress, measured by the PROMIS Pediatric Psychological Stress Experiences 8a | From baseline to post-assessment; approximately 8 weeks
  Youth will report how often (1=never, 5=almost always) they experienced feelings of stress over the past week using the eight-item PROMIS Psychological Stress Experiences-Short Form 8a. As per other PROMIS short forms, summed scores are converted to T-scores.

OTHER OUTCOMES:
Youth Engagement | From baseline to post-assessment, approximately 8 weeks
  The percent of youth who complete at least one activity within the platform, relative to those who complete baseline assessments.
Adverse Childhood Experiences (ACEs) | Baseline
  Youth's lifetime exposure to nine ACEs (e.g., violence, household dysfunction) will be reported by caregivers (if age <18) using items adapted from the National Survey of Children's Health.
Family Demographic Information | Baseline
  Parents/caregivers will report youths' age, sex at birth, racial and ethnic identities, household income, health insurance status/type, and their own highest level of education at baseline.
Youth School Attendance | From baseline to post-assessment; approximately 8 weeks
  Parent/caregivers will report the frequency with which their child misses or is late to school due to physical and/or mental health symptoms over the past month at baseline and after engaging with the self-management platform

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan State University, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
We will not publicly share to protect participant identities but de-identified data may be made available upon reasonable request.